CLINICAL TRIAL: NCT04573621
Title: Pelvic Drain After Rectal Resection for Mid-low Rectal Cancer: a Randomised Controlled Trial
Brief Title: Pelvic Drain After Rectal Resection for Mid-low Rectal Cancer
Acronym: GECO1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GECO1
Record Dates: First submitted 2020-09-24; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessor will not know whether the patient received a drain or not
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic drain (Active Comparator): Placement of a pelvic drain
  Interventions: Procedure: Pelvic drain
- No pelvic drain (Experimental): No pelvic drain placed
  Interventions: Other: No pelvic drain is placed

INTERVENTIONS:
Procedure: Pelvic drain — A pelvic drain is placed
  Arms: Pelvic drain
Other: No pelvic drain is placed — A pelvic drain is not placed
  Arms: No pelvic drain

SUMMARY:
This RCT aims at assessing the effects of a pelvic drain after total mesorectal excision for mid-low rectal cancer on the rates of pelvic sepsis and anastomotic leaks.

DETAILED DESCRIPTION:
This is a 2-arm, non-inferiority RCT. Patients undergoing total mesorectal excision for mid-low rectal cancer will be randomly assigned into two groups:

* pelvic drain
* no pelvic drain. Patients will be followed-up to assess the rates of anastomotic leaks, pelvic sepsis and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, 18 year-of-age or above
* Mid or low rectal cancer
* Anastomosis below the peritoneal reflection
* Total mesorectal excision (TME)
* Capability to understand the study
* Informed consent

Exclusion Criteria:

* For women, pregnancy
* Chronic kidney failure or hepatic failure, immunodepression, malnoutrition
* Life expectancy < 6 months
* Partial mesorectal excision
* Abdominoperineal excision
* Multivisceral resections
* Emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with pelvic sepsis | 0-30 days postoperatively
  anastomotic leak or pelvic collections clinically or radiologically detected

SECONDARY OUTCOMES:
Management of pelvic sepsis | 0-30 days postoperatively
  Type of management (medical, rediological, surgical)
Postoperative complications | 0-30 days postoperatively
  Overall postoperative complications
CT scan or imaging needed | 0-30 days postoperatively
  Necessity of performing unscheduled imaging tests
Number of participants with postoperative ileus | 0-30 days postoperatively
  Postoperative ileus
Diagnostic delay for a leak | 0-30 days postoperatively
  Days between surgery and leak detection
Length of postperative stay | 0-30 days postoperatively or until discharge
  Days of stay after surgery
Time to flatus and bowel movement | 0-30 days postoperatively
  Days between surgery and flatus/faeces
Stoma presence at 1-year follow-up | 12 months after surgery
  Necessity of maintaining the diverting ileostomy at 1-year follow-up
Late pelvic collections | up to 60 days after surgery
  Presence of pelvic collections detected at longer follow-up intervals
Small bowel obstruction | up to 60 days after surgery
  Mechanical small bowel obstruction
Quality of life associated with a drain | 30 days postoperatively
  Visual Analogue Scale 0-10 (higher score means better outcome) score of postoperative pain and wound complaints
Any complications associated with drain removal after surgery | up to 60 days after surgery
  Safety of drain removal after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Universitario Vall d´Hebron, Barcelona, Barcelona, Spain, Spain

IPD SHARING:
Plan to Share IPD: No